CLINICAL TRIAL: NCT00023426
Title: TBTC Study 25:A Prospective, Randomized, Double-Blind Study of the Tolerability of Higher Doses of Rifapentine
Brief Title: TBTC Study 25: Study of the Tolerability of Higher Doses of Rifapentine in the Treatment of Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-2404; HCK45; 25
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2005-09-13 (Estimated); Status verified 2005-09

CONDITIONS: Tuberculosis
Keywords: tuberculosis; tb; rifapentine; safety; dose
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine

INTERVENTIONS:
Drug: rifapentine

SUMMARY:
Randomized, double-blind study of the tolerability of three different doses of rifapentine

DETAILED DESCRIPTION:
Prospective, randomized, double-blinded, comparative study. Patients are randomized at the completion of induction phase therapy. Sample-size is 50 HIV-seronegative patients with culture-positive, drug susceptible TB in each treatment arm. The first 75 patients will be randomized 2:1 to 900 mg:600 mg rifapentine. The second 75 patients will be randomized 2:1 to 1200 mg:600 mg rifapentine. The DSMB will review tolerability and safety data on the first 21 patients enrolled (at the 900 mg and 600 mg doses) and approve proceeding to enrollment at the 1200 mg dose.

ELIGIBILITY:
Inclusions:

1. Drug susceptible culture-positive tuberculosis
2. Adequate induction therapy
3. Age >18
4. Normal screening labs
5. Karnofsky >=60
6. Informed consent
7. Birth control if of child bearing potential

Exclusions:

1. SilicoTB
2. Skeletal or CNS TB
3. Pregnant or breastfeeding
4. Intolerance to INH or rifamycins
5. Over 70 days TB treatment just prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1999-07; Study Completion 2003-02

PRIMARY OUTCOMES:
Proportion of patients who fail to complete therapy in each of the dosing groups

SECONDARY OUTCOMES:
1. Rate of serious adverse events in each of the dosing groups
2. Rate of total adverse events in each of the groups
3. Rate of relapse in patients with positive sputum culture at 2 months, in each of the groups

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Bock, MD, Principal Investigator — Centers for Disease Control & Prevention
Locations (23):
- United States (20):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington, D.C. VAMC, Washington D.C., District of Columbia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nashville VA Medical Center, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Thomas Street Clinic, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec

REFERENCES:
- [Result] Bock NN, Sterling TR, Hamilton CD, Pachucki C, Wang YC, Conwell DS, Mosher A, Samuels M, Vernon A; Tuberculosis Trials Consortium, Centers for Disease Control and Prevention, Atlanta, Georgia. A prospective, randomized, double-blind study of the tolerability of rifapentine 600, 900, and 1,200 mg plus isoniazid in the continuation phase of tuberculosis treatment. Am J Respir Crit Care Med. 2002 Jun 1;165(11):1526-30. doi: 10.1164/rccm.200201-047OC. PMID 12045127
- See also: (Click here for more information about the Tuberculosis Trials Consortium(TBTC) — http://www.cdc.gov/nchstp/tb/tbtc/